CLINICAL TRIAL: NCT06580301
Title: An Open-Label, Multi-Center, Phase Ib/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of YK012 in Participants With B-cell Acute Lymphoblastic Leukemia
Brief Title: Study of YK012 in B-cell Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Excyte Biopharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YK012-2
Record Dates: First submitted 2024-08-26; First posted 2024-08-30 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YK012 (Experimental): Participants will be assigned to a dose level of YK012 based on when the participants join this study.
  Participants will receive YK012 by intravenous infusion (IV), once per week, four weeks per treatment cycle.
  Interventions: Drug: YK012

INTERVENTIONS:
Drug: YK012 — The treatments include 2 cycles of induction treatment, 3 cycles of consolidation treatment, and up to 5 cycles of maintenance treatment.
  Other Names: YK012 for Injection

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics and preliminary anti-tumor activity of YK012 administered as monotherapy in participants with B-cell acute lymphoblastic leukemia (B-ALL).

DETAILED DESCRIPTION:
YK012 is a bispecific antibody designed to link B cells and T cells resulting in T-cell activation and a cytotoxic T-cell response against cluster of differentiation (CD)19 expressing cells. Relapsed/refractory B-ALL in adult patients is an aggressive malignant disease with dismal prognosis. This study is designed in 2 parts as described below: Phase Ib (dose escalation) and Phase II (dose expansion). If in Phase Ib it is observed in adult subjects at doses with manageable risk and antitumor activity, studies in pediatric subjects can be initiated to explore safety and efficacy in pediatric subjects, as well as pharmacokinetic profiles.

ELIGIBILITY:
Inclusion Criteria:

1. Participants or their legally acceptable representative must sign an ICF indicating that the participants understand the purpose of, and procedures required for the study and are willing to participate in the study.
2. Eastern Cooperative Oncology Group Performance Status (ECOG) of 0-2.
3. An estimated survival time of more than 12 weeks.
4. A definitive diagnosis of CD19-positive B-cell acute lymphoblastic leukemia with any of the following conditions:

   1. Ph-negative B-ALL with any of the following: i. Failure to achieve complete remission after initial induction therapy. ii. Failure to achieve complete remission after salvage treatment. iii. Relapse with first remission duration ≤12 months. iv. Second or later relapse. v. Relapse after hematopoietic stem cell transplantation (HSCT).
   2. Ph-positive B-ALL: failure to 1 or more tyrosine kinase inhibitors (TKIs), or intolerance to treatment with TKIs, or with the T315I mutation.
5. ≥ 5% blasts in the bone marrow by morphologic assessment.
6. Recovery to Grade 0-1 (Graded by National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0) from adverse events related to prior therapy except alopecia.
7. Adequate hematological and organ function.
8. Female participants of childbearing potential must have a negative serum pregnancy test at screening. Female patients who are sexually active must use highly effective methods of contraception throughout the study and for 3 months following the last dose of study treatment.
9. Male participants must agree to use reliable methods of contraception (barrier methods or sexual abstinence) and avoid sperm donation throughout the study period and until 3 months after the last dose.

Exclusion Criteria:

1. Burkitt´s Leukemia according to World Health Organization (WHO) classification.
2. History of antitumor therapy as follows, before the first dose of study drug:

   1. Targeted therapy with small molecule drug within 2 weeks or 5 half-lives, whichever is longer
   2. Targeted therapy with macromolecular drug or Immunomodulatory agent therapy within 3 weeks
   3. Radiotherapy or chemotherapy (except for intrathecal chemotherapy and dexamethasone), or treatment with Chinese traditional/patent medicine that has definite antitumor effect within 2 weeks
   4. Treatment with an investigational drug within 4 weeks or 5 half-lives, whichever is shorter
   5. Receipt of any live attenuated vaccines or live virus vaccine within 4 weeks
   6. Autologous stem cell transplantation within 6 weeks
   7. History of organ transplant, or allogeneic stem cell transplantation within 12 weeks.
3. Any active acute graft-versus-host disease (GvHD), grade 2-4 (according to Glucksberg criteria) or active chronic GvHD requiring systemic treatment.
4. Other malignancy within 5 years, except localized malignancies that have been adequately treated or free of the disease for ≥ 5 years, e.g., basal cell carcinoma of the skin, squamous cell carcinoma of the skin, non-muscle invasive bladder cancer, localized prostate cancer, carcinoma in situ of the cervix, carcinoma in situ of the breast.
5. Active central nervous system (CNS) involvement or meningeal involvement with clinical signs, or other evidence of uncontrolled metastases to the CNS or meninges, judged by the investigator.
6. a. History of or current relevant CNS pathology as epilepsy, seizure, paresis, aphasia, apoplexia, severe brain injuries, cerebellar disease, organic brain syndrome, psychosis. b. Evidence for presence of inflammatory lesions and/or vasculitis on cerebral MRI.
7. History or evidence of cardiovascular disease, including:

   1. Acute coronary syndromes (e.g., myocardial infarction, unstable angina)
   2. Coronary angioplasty or stenting within 6 months prior to enrollment
   3. Clinically significant unstable arrhythmias (e.g., atrial fibrillation), however, atrial fibrillation has been controlled for over 30 days prior to the first dose of YK012 were allowed
   4. New York Heart Association (NYHA) stage III or higher congestive heart failure
   5. Left ventricular ejection fraction (LVEF) below lower limit of the study center, or LVEF<50% if there is no lower limit at the study center
   6. The Fridericia-corrected QT interval (QTcF, mean of triplicate measurements) ≥ 470 msec (female) or ≥ 450 msec (male)
   7. Implantable defibrillator
   8. Clinically uncontrollable hypertension (i.e., SBP≥160 mm Hg and/or DBP≥100 mm Hg).
8. Known allergy to monoclonal antibody drugs or exogenous immunoglobulin.
9. History of CD19 targeted therapy and positive test result for immunogenicity of YK012 at screening.
10. Any major organ surgery or significant trauma within 4 weeks prior to the first dose of YK012, or those requiring elective surgeries during the study, and all AEs associated with surgery or significant trauma have not recovered to Grade ≤1 or baseline graded by CTCAE v5.0 before the first dose of the YK012.
11. Regular dose of systemic corticosteroids during 4 weeks prior to initiation of study drug, or anticipated need of corticosteroids exceeding prednisone 20 mg/day or equivalent during the trial, or any other immunosuppressive therapy within 4 weeks prior to study entry.
12. Virological tests: Hepatitis B virus surface antigen (HBsAg) positive and/or hepatitis B core antibody (HBcAb) positive, and hepatitis B virus (HBV) deoxyribonucleic acid (DNA)>ULN of the testing agency; Hepatitis C antibody (HCV-Ab) positive and hepatitis C virus-RNA (HCV-RNA)>ULN of the testing agency; Anti-human immunodeficiency virus (Anti-HIV) positive. Participants will be excluded from the study if any of the above criteria is met.
13. Uncontrolled active infections requiring oral or intravenous systemic therapy, except for local treatment.
14. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage (once a month or more frequently).
15. Pregnant or lactating women.
16. Known mental disorder that may affect study compliance or poor compliance.
17. Other serious systemic diseases or laboratory abnormalities or other reasons that the investigator believes are not appropriate for participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The Incidence and Profile of Dose-limiting Toxicity (DLT) | 28 days after the first dose
  The toxicities occurring within 28 days (i.e., DLT observation period) after the first dose will be defined as DLTs in the discretion of the investigator as related to the IMP (Investigational Medicinal Product).
  This outcome measure is applicable for dose escalation phase only. The MTD dose will be calculated by the statistician upon completion of the dose escalation study.
Maximum Tolerated dose (MTD) or The Recommended Dose for Future Clinical Study | Through study completion, 20 weeks
  This outcome measure is applicable for dose escalation phase only. The MTD dose will be calculated by the statistician upon completion of the dose escalation study.
Number of Participants with Adverse Events | From the time the participant signs the ICF until the end of the safety visit period, assessed up to 24weeks.
  An AE is defined as any untoward medical event that occurs after a subject receives the investigational drug, which may be manifested as symptoms, signs, diseases, or laboratory abnormalities, but may not necessarily have a causal relationship with the investigational drug.
Number of Participants with Serious Adverse Events | From the time the participant signs the ICF until the end of the safety visit period, assessed up to 24weeks.
  An SAE refers to an untoward medical occurrence such as death, life-threatening event, permanent or serious disability or loss of function, need for hospitalization or prolongation of hospitalization after the subject receives the IMP, and congenital abnormalities or birth defects.
Dose Expansion Phase: Objective Response Rate (ORR) | From the time the participant signs the ICF until hematological relapse, assessed up to 1 year
  ORR is defined as percentage of participants achieving either a complete response (CR) or complete remission with partial hematological recovery (CRi).
  The MTD dose will be calculated by the statistician upon completion of the dose escalation study.
  This outcome measure is applicable for dose expansion phase only.

SECONDARY OUTCOMES:
Area Under the Concentration-time Curve (AUC) | Up to 20 weeks
  The PK (AUC) of YK012 will be evaluated.
Maximum Observed Concentration (Cmax) | Up to 20 weeks
  The PK (Cmax) of YK012 will be evaluated.
Time to Reach Maximum Concentration (Tmax) | Up to 20 weeks
  The PK (Tmax) of YK012 will be evaluated.
Half Life (t1/2) of YK012 | Up to 20 weeks
  The PK (t1/2) of YK012 will be evaluated.
Clearance (CL) of YK012 | Up to 20 weeks
  The PK (CL) of YK012 will be evaluated.
Trough Plasma Concentration (Ctrough) | Up to 20 weeks
  The PK (Ctrough) of YK012 will be evaluated.
Percentage of Participants with Anti-Drug Antibody (ADA) and Neutralizing Antibody (Nab) Against YK012 | Up to 20 weeks
  Assess the percentage of participants with ADA and Nab (only assessed when ADA positive except for the screening period) after treatment with YK012.
Dose Escalation Phase: Objective Response Rate (ORR) | From the time the participant signs the ICF until hematological relapse, assessed up to 1 year
  ORR is defined as percentage of participants achieving either a complete response (CR) or complete remission with partial hematological recovery (CRi).
  The MTD dose will be calculated by the statistician upon completion of the dose escalation study.
  This outcome measure is applicable for dose escalation phase only.
Relapse-free Survival (RFS) | From the time the participant signs the ICF until hematological relapse, assessed up to 1 year
  RFS was measured from first dose of YK012 until the first assessment of documented relapse, or death due to any cause, whichever occurs first including the time after the transplant.
Overall survival (OS) | From the date of first dose until loss of follow-up, death, withdrawal of informed consent, or the end of study, whichever occurs first, assessed up to 1 year.
  Overall survival was measured from the first treatment with YK012 until death due to any cause. Participants who did not die were censored at their last contact date.
Number of B cells and T cells in peripheral blood after administration | Up to 20 weeks
  Assess the number of B cells and T cells in peripheral blood after treatment with YK012

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, MD, Principal Investigator — Zhejiang University
Locations (12):
- China (12):
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang